CLINICAL TRIAL: NCT03850158
Title: Visualization of Peritoneal Endometriosis With 2D-Laparoscopy and Indocyanine Green
Brief Title: Diagnostic Value of ICG in Endometriosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Study ID 3300
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Endometriosis; Laparoscopy; Near Infrared Fluorescence Imaging; Indocyanine Green (ICG)
MeSH Terms: conditions — Endometriosis | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Interventional Arm, ICG and NIR imaging (Experimental): NIR fluorescence imaging is performed after white light laparoscopy. 0.3mg/kg bodyweight of ICG is administered i.v. All suspected lesions are removed and labeled whether they are seen in WL or NIR imaging or both. Evaluation is performed after the histological analysis of the lesions.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Indocyanine green is administered intra-venous after dilution with water in a peripheral vein at a dosage of 0.3mg/kg body weight as a bolus injection. The injection will take place during surgery. By using NIR fluorescence imaging ICG is made visible.

SUMMARY:
This study evaluates the diagnostic value of the addition of indocyanine green and near infrared fluorescence imaging during laparoscopy in patients with suspected endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a public health problem with an increasing incidence and various symptoms. Surgical treatment reliefs pain and improves fertility by radically removing endometriotic lesions. However, peritoneal endometriotic lesions may vary significantly in their appearance in standard white light laparoscopy and therefore may be difficult to be identified. Because endometriosis is associated with hypervascularisation the visualization of tissue perfusion by additional use of near infrared (NIR) fluorescence imaging with indocyanine green (ICG) may improve the detection of peritoneal endometriotic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Be premenopausal (menopause is defined as amenorrhea lasting one year or longer)
* Patients should be in follicular phase
* Have chronic pelvic pain and/or Infertility and be willing to undergo planned endometriosis resection procedure.

Exclusion Criteria:

* Known or suspected allergy to iodine, shellfish, or ICG dye
* Hyperthyroidism
* Severe renal insufficiency
* Simultaneous therapy with beta-blockers
* Women who are pregnant (positive HCG in the blood) or breast feeding
* Intention to become pregnant during the course of the study
* Inability to follow the procedures of the study (due to language problems, psychological disorders, dementia)
* Active pelvic infection (positive vaginal or cervical smears for bacteria or elevated markers of infection in the blood)
* Previous history of radiation therapy of the pelvis
* Presence of medical conditions contraindicating general anesthesia or standard laparoscopic surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of detected endometriotic lesions with NIR fluorescence imaging compared to white light laparoscopy | The duration of the participation is from the signature of the informed consent until the end of the hospitalisation, expected to be on average after 2 to 4 days
  The number of histologically proven endometriotic lesions detected with NIR fluorescence imaging are compared to the number of lesions detected with white light laparoscopy alone and white light laparoscopy plus NIR fluorescence imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Imboden, MD, Principal Investigator — Department of Obstetrics and Gynecology, University Hospital of Bern, Inselspital, Switzerland
Locations (1):
- Department of Obstetrics and Gynecology, University Hospital of Bern, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegenthaler F, Knabben L, Mohr S, Nirgianakis K, Imboden S, Mueller MD. Visualization of endometriosis with laparoscopy and near-infrared optics with indocyanine green. Acta Obstet Gynecol Scand. 2020 May;99(5):591-597. doi: 10.1111/aogs.13803. Epub 2020 Jan 28. PMID 31943126